CLINICAL TRIAL: NCT02319278
Title: DEtection of Cellular Inflammation With FERumoxytol in the HEART
Acronym: DECIFER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Royal Infirmary of Edinburgh (Other); Golden Jubilee National Hospital (Other Government); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-002336-24
Record Dates: First submitted 2014-12-03; First posted 2014-12-18 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Cardiac Transplant; Cardiac Sarcoid; Myocarditis; Healthy Volunteers
MeSH Terms: conditions — Myocarditis | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Myocarditis (Active Comparator)
  Interventions: Drug: Ferumoxytol
- Cardiac sarcoid (Active Comparator)
  Interventions: Drug: Ferumoxytol
- Cardiac Transplant (Active Comparator)
  Interventions: Drug: Ferumoxytol
- Healthy Volunteers (Placebo Comparator)
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — Infusion following between paired MRI scans

SUMMARY:
To non-invasively image myocardial accumulation of ultrasmall superparamagnetic particles of iron oxide (USPIOs) by an increase in R2* values (compared to controls) within the myocardium of patients with:

i. cardiac transplantation ii. acute myocarditis iii. suspected cardiac sarcoidosis

DETAILED DESCRIPTION:
Ferumoxytol is a 'smart' magnetic resonance contrast agent consisting of ultrasmall superparamagnetic particles of iron oxide (USPIOs) that are taken up by macrophages. Concentration of USPIOs within macrophages changes the tissue relaxation properties and this can be detected by magnetic resonance imaging using R2* maps. In a recent early proof-of-concept study, we demonstrated that macrophages could be detected with USPIOs in the penumbra and infarct zone of the myocardium in patients with a recent myocardial infarction. The investigators therefore wish to establish whether USPIOs can be used to identify cellular inflammation within the myocardium in three distinct clinical conditions that currently lack a non-invasive diagnostic imaging test: cardiac allograft rejection, viral myocarditis and cardiac sarcoidosis. If successful, this would not only provide a useful diagnostic test but would also be a method of monitoring disease progression or response to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. One of the four conditions below:

   * Patients having undergone cardiac transplant
   * Patients diagnosed clinically with myocarditis of any aetiology (eg viral, septic, post chemotherapeutic etc)
   * Patients clinically diagnosed with cardiac sarcoidosis
   * Healthy volunteers
2. Age > 18 years.

Exclusion Criteria:

1. Contraindication to magnetic resonance imaging scanning identified from magnetic resonance imaging safety questionnaire
2. Patients refusing or unable to give informed consent
3. Renal failure (estimated glomerular filtration rate <30 mL/min)
4. Polycythemia
5. Contraindication to ferumoxytol (previous allergic drug reaction, any immune or inflammatory conditions (eg, systemic lupus erythematosus, rheumatoid arthritis, history of severe asthma, eczema or other atopic allergy)), evidence of known iron overload, hemochromatosis, known hypersensitivity to ferumoxytol or its components or anaemia not caused by iron deficiency.
6. Known allergy to dextran- or iron-containing compounds.
7. Diagnosis of myocardial infarction within 1 month.
8. Pregnancy or Breast-feeding.
9. Women of child bearing age not ensuring reliable methods of contraception. Female participants of child bearing age will be asked if they are ensuring reliable methods of contraception prior to each administration of USPIO and MRI scan. If use of reliable contraception cannot be confirmed, the participant will be withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Myocardial Cellular Inflammation. | 1 year
  Assessment of Myocardial Cellular Inflammation through the increase in R2* value on post USPIO imaging versus baseline imaging.

SECONDARY OUTCOMES:
Correlation of R2* values with circulating inflammatory markers | 1 year
  Comparison of circulating inflammatory markers in peripheral blood with myocardial inflammation (seen on cardiac R2* maps) .
Does clinical condition correlate with inflammation seen on R2* maps. (assessed by reduction in R2* values) | 1 year
  Does treatment or recovery from these inflammatory myocardial conditions reduce or halt uptake of USPIOs as assessed by reduction in R2* values.
Do higher R2* correlate with poorer outcome? (assessed by deterioration in ejection fraction or increase in late gadolinium enhancement) | 1 year
  Do patients with higher R2* values have worse outcomes assessed by deterioration in ejection fraction or increase in late gadolinium enhancement.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Stirrat, MBChB, Principal Investigator — University of Edinburgh
Locations (3):
- United Kingdom (3):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Golden Jubilee National Hospital, Glasgow
  - Royal Brompton Hospital, London

REFERENCES:
- [Derived] Stirrat CG, Alam S, MacGillivray TJ, Gray C, Dweck MR, Jones V, Wallace W, Payne JR, Prasad SK, Gardner RS, Petrie MC, Mirsadraee S, Henriksen P, Newby DE, Semple S. Ferumoxytol-enhanced MRI in patients with prior cardiac transplantation. Open Heart. 2019 Oct 3;6(2):e001115. doi: 10.1136/openhrt-2019-001115. eCollection 2019. PMID 31673393
- [Derived] Stirrat CG, Alam SR, MacGillivray TJ, Gray CD, Dweck MR, Dibb K, Spath N, Payne JR, Prasad SK, Gardner RS, Mirsadraee S, Henriksen PA, Semple SI, Newby DE. Ferumoxytol-enhanced magnetic resonance imaging in acute myocarditis. Heart. 2018 Feb;104(4):300-305. doi: 10.1136/heartjnl-2017-311688. Epub 2017 Oct 6. PMID 28986407
- [Derived] Stirrat CG, Alam SR, MacGillivray TJ, Gray CD, Dweck MR, Raftis J, Jenkins WS, Wallace WA, Pessotto R, Lim KH, Mirsadraee S, Henriksen PA, Semple SI, Newby DE. Ferumoxytol-enhanced magnetic resonance imaging assessing inflammation after myocardial infarction. Heart. 2017 Oct;103(19):1528-1535. doi: 10.1136/heartjnl-2016-311018. Epub 2017 Jun 22. PMID 28642288
- [Derived] Stirrat CG, Alam SR, MacGillivray TJ, Gray CD, Forsythe R, Dweck MR, Payne JR, Prasad SK, Petrie MC, Gardner RS, Mirsadraee S, Henriksen PA, Newby DE, Semple SI. Ferumoxytol-enhanced magnetic resonance imaging methodology and normal values at 1.5 and 3T. J Cardiovasc Magn Reson. 2016 Jul 27;18(1):46. doi: 10.1186/s12968-016-0261-2. PMID 27465647